CLINICAL TRIAL: NCT07126080
Title: The Effect of Coping Training on Urinary Incontinence Attitudes, Sleep, and Quality of Life in Postmenopausal Women With Stress Urinary Incontinence: A Randomized Controlled Trial
Brief Title: Effect of Coping Training on Attitudes, Sleep, and Quality of Life in Women With Stress Urinary Incontinence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Dilek Celi̇k Eren, Ass. Prof., Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2025-845; There is no funding. (Other: Researchers will carry out this with their own budget.)
Record Dates: First submitted 2025-07-29; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Stress Urinary Incontinence
Keywords: Postmenopausal; Stress Urinary Incontinence; coping strategies; health quality; Attitude; Sleep Quality
MeSH Terms: conditions — Urinary Incontinence, Stress; Behavior; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: randomized controlled pretest-posttest control group experimental research design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group-Training in Coping with Incontinence (Experimental): Intervention: Women in the experimental group will receive a four-week training program on managing urinary incontinence. The training will cover the following topics:
  * Definition, types, and risk factors of urinary incontinence
  * Treatment and prevention of urinary incontinence
  * Symptoms of urinary incontinence and non-drug management strategies (addressing eating and toilet habits, such as limiting caffeinated beverages and cautioning spicy foods)
  * The importance and implementation of Kegel exercises After the training, the experimental group will be reminded to practice Kegel exercises, and post-tests will be administered at 1 and 3 months. The control group will also receive post-tests at 1 and 3 months. Training will be conducted individually online.
  Interventions: Behavioral: Incontinence Coping Training
- Control Group (No Intervention): No ıntervention.

INTERVENTIONS:
Behavioral: Incontinence Coping Training — Intervention: Women in the experimental group will receive a four-week training program on managing urinary incontinence. The training will cover the following topics:
  * Definition, types, and risk factors of urinary incontinence
  * Treatment and prevention of urinary incontinence
  * Symptoms of urinary incontinence and non-drug management strategies (addressing eating and toilet habits, such as limiting caffeinated beverages and cautioning spicy foods)
  * The importance and implementation of Kegel exercises After the training, the experimental group will be reminded to practice Kegel exercises, and post-tests will be administered at 1 and 3 months. The control group will also receive post-tests at 1 and 3 months. Training will be conducted individually online.
  Arms: Intervention Group-Training in Coping with Incontinence

SUMMARY:
This study aims to examine the effects of urinary incontinence management training provided to postmenopausal women on their urinary incontinence attitudes, sleep, and quality of life.

Hypothesis H1: Following the urinary incontinence management training, there will be an increase in urinary incontinence attitudes, sleep, and quality of life in the women in the experimental group compared to the women in the control group.

DETAILED DESCRIPTION:
1. Research Model: This study will be conducted using a randomized controlled pretest-posttest control group experimental research design.
2. Research Universe/Sample or Study Group:

   This study will be conducted with postmenopausal women over the age of 45 who attended the Gynecology and Obstetrics Clinic of Ondokuz Mayıs University Health Application and Research Center. The study sample size was calculated using the sample size calculator program. Using the Urinary Incontinence Quality of Life Scale as a reference (12.34 (2.18); 5.43 (1.96)) (Başgöl et al., 2025), the sample size was calculated as 36 participants for the experimental group and 36 participants for the control group, with a 5% margin of error, a 90% confidence interval, and an effect size of 33.332. In addition to the minimum sample size, a sample size of 48 participants was determined for each group, with at least 50% spares, for a total of 96 participants. Randomization Simple randomization will be used to unbiasedly assign 96 women who meet the study criteria to the intervention and control groups. Randomization will be determined computer-aided using the Research Randomizer website (https://www.randomizer.org/). Women in the intervention and control groups will be assigned based on the obtained order.
3. Data Collection Tools: A Personal Information Form, the Urinary Incontinence Short Test, the Pittsburgh Sleep Quality Index, and the Urinary Incontinence Quality of Life Scale (I-QOL) will be used to collect data for the study.

   Personal Information Form: Consists of a total of 21 questions that ask about the women's sociodemographic characteristics such as age, education level, and income, their characteristics related to childbirth, and their experience of urinary incontinence. Urinary Incontinence Attitude Scale:

   Pittsburg Sleep Quality Index: The scale's validity and reliability studies in Turkey were conducted by Ağargün and colleagues in 1996. The PSQI assesses sleep quality over the past month. The PSQI consists of 24 questions, 19 of which are answered by the individual themselves, and 5 by their spouse or roommate. The total score ranges from 0 to 21. A high total score indicates poor sleep quality. A total PSQI score greater than 5 is considered the cut-off score indicating poor sleep quality. The scale's Cronbach's alpha reliability coefficient was found to be 0.804.

   Urinary Incontinence Quality of Life Scale (I-QOL): The validity and reliability of the I-QOL was performed by Özerdoğan. In the Incontinence Quality of Life Scale, all items are evaluated on a five-item Likert-type scale (1=a lot, 2=quite a bit, 3=moderately, 4=a little, 5=not at all), and the calculated total score is converted to a scale value from 0 to 100 for better understanding. The Incontinence Quality of Life Scale consists of three subscales: restrictive behaviors (items 1, 2, 3, 4, 10, 11, 13, and 20), psychological impact (items 5, 6, 7, 9, 15, 16, 17, 21, and 22), and limitations on social life (items 8, 12, 14, 18, and 19). Higher scores indicate better quality of life than lower scores.

   Incontinence Short Test: To determine the level of knowledge about incontinence, Branch et al. The Incontinence Short Test, developed by Kara et al. and whose Turkish version was studied by Kara et al., was used. The 14-item test is answered with "Agree," "Disagree," or "Don't Know." The correct answer for items 1, 4, 6, 8, 10, and 11 is "Agree." For the remaining items, the correct answer is "Disagree." A "Don't Know" response is considered incorrect. The total score ranges from 0 to 14, with a higher score indicating a higher level of knowledge and a more positive attitude toward urinary incontinence.

   Intervention: The women in the experimental group will receive a 4-week training program on coping with urinary incontinence. The content of this training consists of the following topics: • Definition, types, and risk factors for urinary incontinence
   * Treatment and prevention of urinary incontinence
   * Non-drug management strategies for managing urinary incontinence symptoms (eating and toilet habits, such as limiting caffeinated beverages and being mindful of spicy foods)
   * Importance and implementation of Kegel exercises After the training is completed, the experimental group will be reminded to practice Kegel exercises, and post-tests will be administered at 1 and 3 months. The control group will also be given post-tests at 1 and 3 months. Training will be conducted individually via an online platform.
4. Data Collection Process: Pre-tests will be administered to the women in the experimental and control groups at the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Having entered menopause
* Volunteering to participate in the study
* Having no communication barriers
* Using a smartphone
* Having the WhatsApp application
* Experiencing urine leakage when coughing or sneezing, as defined by the ICS (International Continence Association)

Exclusion Criteria:

* Having a communication barrier
* Not having gone through menopause
* Not experiencing urinary incontinence
* Having undergone surgical menopause
* Being obese

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 96 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Personal Information Form | 4 weeks
  It consists of a total of 21 questions asking about women's sociodemographic characteristics such as age, education level, income level, birth-related characteristics and urinary incontinence.
The incontinence short test: | 16 weeks
  A Turkish validity and reliability study was conducted by Kara et al. The test consists of 14 statements and is answered with "Agree," "Disagree," or "Don't Know." The correct answer for statements 1, 4, 6, 8, 10, and 11 is "Agree." The correct answer for the remaining statements is "Disagree." A "Don't Know" response is considered incorrect. The total score ranges from 0 to 14, with higher scores indicating a higher level of knowledge and a more positive attitude toward urinary incontinence.
Pittsburgh Sleep Quality Index: | 16 weeks
  The scale's validity and reliability studies in Turkey were conducted by Ağargün and colleagues in 1996. The PSQI assesses sleep quality over the past month. The PSQI consists of 24 questions, 19 of which are answered by the individual themselves, and 5 by their spouse or roommate. The total score ranges from 0 to 21. A high total score indicates poor sleep quality. A total PSQI score of 5 or higher is considered the cut-off score for poor sleep quality. The scale's Cronbach's alpha reliability coefficient was found to be 0.804.
Urinary Incontinence Quality of Life Scale (I-QOL): | 16 weeks
  The validity and reliability of the I-QOL was determined by Özerdoğan. All items in the Incontinence Quality of Life Scale are evaluated on a five-category Likert-type scale (1=a great deal, 2=quite a bit, 3=moderately, 4=a little, 5=not at all), and the calculated total score is converted to a scale value from 0 to 100 for better understanding. The Incontinence Quality of Life Scale consists of three subscales: behavioral limitation (items 1, 2, 3, 4, 10, 11, 13, and 20), psychological impact (items 5, 6, 7, 9, 15, 16, 17, 21, and 22), and social limitation (items 8, 12, 14, 18, and 19). High scores indicate better quality of life than low scores.
Personal Information Form | 16 weeks
  It consists of a total of 21 questions asking about women's sociodemographic characteristics such as age, education level, income level, birth-related characteristics and urinary incontinence.

CONTACTS AND LOCATIONS:
Overall Officials: İlknur AYDIN AVCİ, Prof. Dr., Study Director — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs University, Samsun, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided